CLINICAL TRIAL: NCT01248663
Title: Influence of the Reconstruction Method on the Incidence of Delayed Gastric Emptying After Pylorus Preserving Pancreaticoduodenectomy. A Prospective, Randomized Trial.
Brief Title: Reconstruction Method and Delayed Gastric Emptying After Pancreatic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Michael Gnant, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-020
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer; Surgery; Improvement of Perioperative Outcome
Keywords: pancreatic cancer; pylorus-preserving pancreaticoduodenectomy; delayed gastric emptying; reconstruction
MeSH Terms: conditions — Pancreatic Neoplasms; Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- antecolic reconstruction (Active Comparator): After completion of pancreaticoduodenectomy and reconstruction of the pancreaticojejunostomy and hepaticojejunostomy, the reconstruction of the intestinal passage will be conducted by performing an antecolic duodeno-jejunostomy
  Interventions: Procedure: antecolic reconstruction
- retrocolic reconstruction (Experimental): After completion of pancreaticoduodenectomy and reconstruction of the pancreaticojejunostomy and hepaticojejunostomy, the reconstruction of the intestinal passage will be conducted by performing a retrocolic duodeno-jejunostomy
  Interventions: Procedure: retrocolic reconstruction

INTERVENTIONS:
Procedure: antecolic reconstruction — see study arm description
  Arms: antecolic reconstruction
Procedure: retrocolic reconstruction — see study arm description
  Arms: retrocolic reconstruction

SUMMARY:
Pancreaticoduodenectomy (whipple procedure) is the standard operation for tumors of the pancreatic head, uncinate process, distal common bile duct as well as the papilla of vater. For reconstruction, pylorus-preservation (PPPD) has been shown to be technically and oncologically equivalent to the traditional whipple operation. One issue with this technique is delayed gastric emptying (DGE), which occurs in 25-70% of patients, usually emerging between day 4 and 14 after surgery. Patients with severe DGE can not only experience prolonged length of hospital stay, but are also at increased risk for other complications like aspiration or other issues related to the inability to ingest nutrition.

There is vast retrospective evidence and one prospective study indicating that antecolic reconstruction of the duodenojejunostomy can improve the rate and severity of delayed gastric emptying.

The investigators have conducted a prospective randomized trial in order to test this hypothesis. Patients were randomized to either undergo antecolic or retrocolic reconstruction after PPPD. On day 10 after surgery, DGE was assessed by clinical criteria. In addition, a test meal including 1g paracetamol was administered to check for clinically inapparent DGE. Of these serum samples, kinetics of intestinal peptides like GLP-1, PYY and glucagon was alos measured.

ELIGIBILITY:
Inclusion Criteria:

* verified cancer of the pancreatic head/neck/uncinate process or distal bile duct, radiographically suspicious tumor requiring pancreaticoduodenectomy
* pylorus-preserving reconstruction planned
* no evidence of distant metastases
* written informed consent

Exclusion Criteria:

* age <18 or >90 years
* status post surgical resection of stomach or duodenum
* locally unresectable:
* invasion of the hepatic artery/superior mesenteric artery
* >180 deg invasion of portal vein/superior mesenteric vein
* gastric invasion
* hypersensitivity to paracetamol
* clinically significant anastomotic dehiscence
* postoperative pancreatitis > day 10
* preoperative evidence of gastroparesis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Delayed gastric emptying | Postoperative day 10
  Gastric emptying will be assessed by clinical criteria on postoperative day 10 after pylorus-preserving pancreatico-duodenectomy.

SECONDARY OUTCOMES:
Paracetamol reabsorption test | postoperative day 10
  On day 10 after pylorus-preserving pancreaticoduodenectomy, a test meal of a commercially available dietary product (Fresubin protein energy(c)) and 1g paracetamol will be administered. Serum levels of paracetamol will be measured at 0, 15, 30, 60 and 90 minutes after administration.
Measurement of plasma intestinal peptides | postoperative day 10
  On day 10 after pylorus-preserving pancreaticoduodenectomy, a test meal of a commercially available dietary product (Fresubin protein energy(c)) and 1g paracetamol will be administered. Serum levels of glucagon-like peptide-1 (GLP-1), peptide YY (PYY) and Glucagon will be measured at 0, 15, 30, 60 and 90 minutes after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gnant, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria